CLINICAL TRIAL: NCT04312633
Title: CDx Study 906: The Clinical Utility of WATS3D (Wide Area Transepithelial Sampling With Computer-Assisted 3-Dimensional Analysis): A 5- Year Prospective Registry
Brief Title: Clinical Utility of WATS3D: A 5-Year Prospective Study
Status: Recruiting | Type: Observational
Sponsor: CDx Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CDx 906
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Barrett Esophagus; Gastro Esophageal Reflux; Esophageal Dysplasia; Esophageal Diseases
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Esophageal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to create a registry (collect data and keep it in a research database) to learn more about two methods of taking small tissue samples from your esophagus (the esophagus is the tube that carries food and liquid from your mouth to your stomach). The two methods of sampling are: 1) Using forceps that take biopsies (small tissue samples) from your esophagus, and 2) Using a brush that also takes biopsies from your esophagus.

DETAILED DESCRIPTION:
This study will look at the impact of the brush biopsy results on your doctor's decisions about your future care and treatment.

In addition , by recording the results of all your biopsies over 5 years, it may be possible to find out if the brush biopsy, forceps biopsy, or both can predict which patients with heartburn develop Barrett's esophagus, (an abnormality in the esophagus that may lead to cancer), and which patients with Barrett's esophagus develop precancer and cancer.

You are being asked to participate in the study because you are receiving an upper endoscopy (a procedure where a tube with a light and camera are inserted in your mouth and down your throat) with forceps and brush biopsies of your esophagus as part of you standard clinical care, and you are at least 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, comprehend and complete the IRB-approved consent form
* Aged 18 or older
* Meet one of the following:
* Patients with heartburn or regurgitation undergoing a screening EGD, who undergo WATS3D sampling and forceps biopsies for suspicion of BE, or
* Patients with known BE with or without dysplasia undergoing a surveillance EGD with WATS3D biopsies and forceps biopsies, or
* Patients who have undergone endoscopic eradication (i.e. radiofrequency ablation or cryoablation) who are undergoing surveillance EGD following the establishment of complete eradication of intestinal metaplasia (CEIM)
* Only patients who undergo both forceps biopsies and WATS3D of the esophagus will be included.

Exclusion Criteria:

* Pregnancy at time of endoscopy
* Unresolved drug or alcohol dependency that will limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions or follow-up guidelines
* Medical condition that will likely prohibit completion of a 5 year study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with heartburn or regurgitation undergoing a screening EGD, who undergo WATS3D sampling and forceps biopsies for suspicion of BE, or
  * Patients with known BE with or without dysplasia undergoing a surveillance EGD with WATS3D biopsies and forceps biopsies, or
  * Patients who have undergone endoscopic eradication (i.e. radiofrequency ablation or cryoablation) who are undergoing surveillance EGD following the establishment of complete eradication of intestinal metaplasia (CEIM)
Sampling Method: Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: | 5 years
  Clinical Utility of WATS3D as determined by how many patients undergo increased surveillance, radiofrequency ablation and placement on PPIs.

SECONDARY OUTCOMES:
Secondary Outcome Measure: | 5 years
  Incremental detection yield due to WATS sampling as number of patients who have Barrett's Esophagus and Esophageal Dysplasia determined by WATS and missed by forceps biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew McKinley, M.D., Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Ambulatory Care, Bethpage, New York, United States